CLINICAL TRIAL: NCT01047007
Title: A Phase I Dose Escalation Study of MK1775 in Monotherapy, in Combination With 5-Fluorouracil, and in Combination With 5-Fluorouracil and Cisplatin in Patients With Advanced Solid Tumor
Brief Title: A Dose Escalation Study of Adavosertib(MK1775) in Combination With 5-FU or 5-FU/CDDP in Patients With Advanced Solid Tumor (1775-005
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated due to business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1775-005; MK1775-005 (Other: Merck Registration Number)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors
Keywords: Head and Neck Cancer; Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — adavosertib; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: adavosertib 65 mg BID (Experimental): Participants received 65 mg of adavosertib administered orally twice a day (BID) on Days 1-5 of a 21-day cycle.
  Interventions: Drug: adavosertib 65 mg
- Part 2 A1: adavosertib 20 mg BID+5-FU 1000 mg (Experimental): Participants received 20 mg of adavosertib administered orally BID on Days 1-5 of a 21-day cycle and 1000 mg/m^2/day of 5-FU administered as an intravenous (IV) infusion on Days 1-4 of a 21-day cycle.
  Interventions: Drug: adavosertib 20 mg; Drug: 5-FU 1000 mg/m^2/day
- Part 2 A2: adavosertib 20 mg QD+5-FU 1000 mg (Experimental): Participants received 20 mg of adavosertib administered orally once a day (QD) on Days 1-5 of a 21-day cycle and 1000 mg/m^2/day of 5-FU administered as an IV infusion on Days 1-4 of a 21-day cycle.
  Interventions: Drug: adavosertib 20 mg; Drug: 5-FU 1000 mg/m^2/day
- Parts 2B +3: adavosertib+5-FU+CDDP (Experimental): Participants were to receive 20 mg or 65 mg of adavosertib administered either BID or QD on Days 1-5 of a 21-day cycle; 1000 mg/m^2/day of 5-FU administered as an IV infusion on Days 1-4 of a 21-day cycle; and 60 mg/m^2 to 100 mg/m^2 of CDDP administered as an IV infusion on Day 1.
  Interventions: Drug: adavosertib 20 mg; Drug: 5-FU 1000 mg/m^2/day; Drug: CDDP; Drug: adavosertib 65 mg

INTERVENTIONS:
Drug: adavosertib 20 mg — Adavosertib 20 mg capsule administered orally on days 1-5 of a 21 day cycle.
  Other Names: MK-1775
  Arms: Part 2 A1: adavosertib 20 mg BID+5-FU 1000 mg; Part 2 A2: adavosertib 20 mg QD+5-FU 1000 mg; Parts 2B +3: adavosertib+5-FU+CDDP
Drug: 5-FU 1000 mg/m^2/day — 5-FU 1000 mg/m^2/day administered as an intravenous (IV) infusion on Days 1-4 of a 21-day cycle
  Arms: Part 2 A1: adavosertib 20 mg BID+5-FU 1000 mg; Part 2 A2: adavosertib 20 mg QD+5-FU 1000 mg; Parts 2B +3: adavosertib+5-FU+CDDP
Drug: CDDP — CDDP 60 mg/m^2 to 100 mg/m^2 administered as an IV infusion on Day 1.
  Other Names: Cisplatin
  Arms: Parts 2B +3: adavosertib+5-FU+CDDP
Drug: adavosertib 65 mg — Adavosertib 65 mg capsule administered orally on days 1-5 of a 21 day cycle.
  Other Names: MK-1775
  Arms: Part 1: adavosertib 65 mg BID; Parts 2B +3: adavosertib+5-FU+CDDP

SUMMARY:
The study evaluates safety of adavosertib in monotherapy, and in combination with 5-Fluorouracil (5-FU) alone or with 5-FU/cis-diamminedichloroplatinum (CDDP) in Japanese participants with solid tumor. The primary hypothesis is that adavosertib is safe and tolerable in participants with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Parts 1 and 2-A: Patient must have a histologically or cytologically confirmed locally advanced or metastatic solid tumor failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist
* Parts 2-B and 3: Patient must have a histologically or cytologically confirmed locally advanced or metastatic esophageal, head and neck, or gastric cancer, and be a candidate of 5-Fluorouracil and Cisplatin regimen defined in this study
* Patient must have performance status of 0 or 1 on the ECOG Performance Scale

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy, or biological therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first dose of study drug or who has not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patient with a known primary central nervous system tumor
* Patient has known hypersensitivity to any of the components of the combination study therapy or its analogs
* Patient is receiving "alternative" cancer medications such as plant-derived products and their analogs with anti-tumor activity within 1 week prior to entering the study.
* Patient must not have prior radiation therapy to more than 30% of the bone marrow and must have recovered for at least 3 weeks from the hematologic toxicity of prior radiotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01-18 (Actual); Primary Completion 2011-06-15 (Actual); Study Completion 2011-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with a confirmed locally advanced or metastatic solid tumor failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Additional inclusion and exclusion criteria applied.
Pre-assignment Details: Participants received MK-1775 (Part 1), MK-1775 + 5-Fluorouracil (Part 2A), and MK-1775 + 5-Fluorouracil and cis-diamminedichloroplatinum (Parts 2B and 3). The study was terminated early and Parts 2B and 3 were not performed. No participants received the 5-Fluorouracil (5-FU) and cis-diamminedichloroplatinum (CDDP) regimen.
Groups:
- Part 1: MK-1775 65 mg BID: Participants received 65 mg of MK-1775 administered orally twice a day (BID) on Days 1-5 of a 21-day cycle.
- Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg: Participants received 20 mg of MK-1775 administered orally BID on Days 1-5 of a 21-day cycle and 1000 mg/m^2/day of 5-FU administered as an intravenous (IV) infusion on Days 1-4 of a 21-day cycle.
- Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg: Participants received 20 mg of MK-1775 administered orally once a day (QD) on Days 1-5 of a 21-day cycle and 1000 mg/m^2/day of 5-FU administered as an IV infusion on Days 1-4 of a 21-day cycle.
- Parts 2B +3: MK-1775 + 5-FU + CDDP: Participants were to receive 20 mg or 65 mg of MK-1775 administered either BID or QD on Days 1-5 of a 21-day cycle; 1000 mg/m^2/day of 5-FU administered as an IV infusion on Days 1-4 of a 21-day cycle; and 60 mg/m^2 to 100 mg/m^2 of CDDP administered as an IV infusion on Day 1.
Period: Overall Study
Arm/Group | Part 1: MK-1775 65 mg BID | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg | Parts 2B +3: MK-1775 + 5-FU + CDDP
Started | 3 | 6 | 2 | 0
Treated | 3 | 6 | 2 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 2 | 6 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Progressive Disease | 2 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-1775 65 mg BID | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg | Parts 2B +3: MK-1775 + 5-FU + CDDP | Total
Number analyzed (Participants) | 3 | 6 | 2 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (4.4) | 62.7 (7.9) | 59.0 (5.7) |  | 62.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 |  | 1
  Male | 3 | 5 | 2 |  | 10
ECOG Performance Status [Number; unit: Participants] — The ECOG scale of performance status is a measurement of how the disease impacts the daily living abilities of the participant. It describes a participant's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. The scale ranges from 0 (fully active) to 5 (dead). The study required participants to have a score of 0 (fully active, able to carry on all pre-disease performance without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG Score = 0 | 2 | 3 | 2 |  | 7
    ECOG Score = 1 | 1 | 3 | 0 |  | 4
Number of Prior Chemotherapy Regimens [Mean (Standard Deviation); unit: Prior regimens] — The study required participants to have a solid tumor that failed to respond to standard therapy or progressed despite standard therapy as demonstrated by the number of prior chemotherapy regimens received.
  Prior regimens | 2.0 (0.0) | 3.3 (0.8) | 4.0 (0.0) |  | 3.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined using National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 and included: any drug-related hematologic toxicity ≥Grade 4 with the exception of Grade 4 neutropenia <7 days duration; Grade 3 or 4 neutropenia with fever >38.5 degrees Celsius and/or infection or neutropenia requiring colony-stimulating factor OR non-hematologic DLTs that were any Grade 3, 4, or 5 toxicity with the following exceptions: Grade 3 nausea, vomiting, diarrhea, and dehydration occurring in a setting of inadequate treatment; inadequately treated hypersensitivity reactions; Grade 3 elevated transaminases or urine electrolyte abnormality ≤1 week in duration; Grade 3 serum electrolyte abnormality ≤72 hours in duration. DLTs also included: drug-related adverse experience that lead to a dose modification; unresolved drug-related toxicity preventing treatment for ≥3 weeks or preventing administration of ≥8 of 10 doses in Parts 1 or 2A1 or 4 of 5 doses in Part 2A2.
Time Frame: Cycle 1 (21 days)
Population: The DLT-evaluable population consisted of participants who received at least one dose of MK-1775 and completed Cycle 1 of Parts 1, 2A1, 2A2, or discontinued due to toxicity.
Measure: Number; unit: Participants
Arm/Group | Part 1: MK-1775 65 mg BID | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg | Parts 2B +3: MK-1775 + 5-FU + CDDP
Number analyzed (Participants) | 3 | 6 | 2 | 0
Participants | 0 | 1 | 1 |

2. Primary Outcome: Maximum Tolerated Dose (MTD) of MK1775 in Combination With 5-FU/CDDP Determined by Number of DLTs Per Dose Level: Locally Advanced or Metastatic Esophageal, Head and Neck, or Gastric Cancer
Description: The maximum tolerated dose (MTD) of MK-1775 in combination with 5-FU/CDDP for participants with locally advanced or metastatic esophageal, head and neck, or gastric cancer was determined based on DLTs that occurred during Cycle 1 of Parts 2B and 3. The MTD for MK-1775 in combination with 5-FU/CDDP was defined as the dose level at which approximately 30% of the participants were expected to experience a DLT for the combination therapy. The study was terminated early and Parts 2B and 3 were not performed. No participants received the 5-FU/CDDP regimen therefore the MTD for MK-1775 in combination with 5-FU/CDDP was not established.
Time Frame: Cycle 1 (21 days)
Population: Participants who received at least one dose of MK-1775 in combination with 5-FU/CDDP and completed Cycle 1 of Parts 2B and 3. No participants received the 5-FU/CDDP regimen due to early termination of the study.
Arm/Group | Parts 2B +3: MK-1775 + 5-FU + CDDP
Number analyzed (Participants) | 0

3. Secondary Outcome: MTD of MK1775 in Combination With 5-FU/CDDP Determined by Number of DLTs Per Dose Level: Locally Advanced or Metastatic Solid Tumors
Description: The maximum tolerated dose (MTD) of MK-1775 in combination with 5-FU/CDDP for participants with locally advanced or metastatic solid tumors was determined based on DLTs that occurred during Cycle 1 of Parts 2B and 3. The MTD for MK-1775 in combination with 5-FU/CDDP was defined as the dose level at which approximately 30% of the participants were expected to experience a DLT for the combination therapy. The study was terminated early and Parts 2B and 3 were not performed. No participants received the 5-FU/CDDP regimen therefore the MTD for MK-1775 in combination with 5-FU/CDDP was not established.
Time Frame: Cycle 1 (21 days)
Population: as for outcome 2
Arm/Group | Parts 2B +3: MK-1775 + 5-FU + CDDP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of MK-1775 alone or in combination with 5-FU through follow-up; up to 7 months
Description: AEs for all participants who received at least one dose of MK-1775 alone or in combination with 5-FU.
Arm/Group | Part 1: MK-1775 65 mg BID | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 65 mg BID (N=3) | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg (N=6) | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg (N=2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 65 mg BID (N=3) | Part 2 A1: MK-1775 20 mg BID + 5-FU 1000 mg (N=6) | Part 2 A2: MK-1775 20 mg QD + 5-FU 1000 mg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (8) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (7) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (5) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 2 (5) | 3 (9) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (11) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (5) | 1 (2)
Infusion site extravasation (General disorders) | 1 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (4) | 0 (0)
Electrocardiogram ST-T segment depression (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to business reasons. Study Parts 2B and 3 were not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.